CLINICAL TRIAL: NCT00577811
Title: Evaluation of Enrollment, Dynamics of Care and Patient Outcomes in the NYS Medicaid HIV Special Needs Plans
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Bruce Rapkin, Ph.D., Memorial Sloan-Kettering Cancer Center
Other Study IDs: 03-011
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections; Mental Health
Keywords: Special Need Plans; Fee for Services; Access to Care; Medicaid
MeSH Terms: conditions — HIV Infections; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients from 6 different Special Need Plans
- 2

SUMMARY:
The purpose of this study is to find out how people's needs are being met and what people do about problems with treatment, symptoms, substance use, mental health, and social services. We are also interested in finding out about changes that people make in their health care team and the reasons for making those changes.

DETAILED DESCRIPTION:
This is a longitudinal study to examine access to care, perceived quality of life, member satisfaction and patient-reported outcomes among HIV+ adult Medicaid recipients. Special Needs Plans represent a new approach to managed care tailored to patients with complicated medical and psychosocial problems,requiring a high level of service. These plans combine HIV primary and specialty care, mental health services, substance use treatment, care for dependent children and social services into a single comprehensive program that also includes comprehensive case management and other provisions to retain patients in care. Special Needs Plans represent an alternative to both, Medicaid Fee for Service (FFS) and to mainstream Medicaid managed care.Seven different Special Needs Plans will be implemented, serving in New York City and the surrounding suburbs. A separate non-profit corporation administers each SpecialNeeds Plan. Each plan encompasses a network of hospitals, providers, and communitybased organizations. Although all plans offer many of the same basic services, they differ in terms of organization and coordination of care, approaches to case management,specific program enhancements (e.g., patient education, wellness programs, or complementary medicine) and special provisions to meet the needs of subgroups of patients (e.g., women, substance users, young gay men, Latinos). The HIV Special Needs Plans represent an innovation in health service delivery and financing that is being evaluated as a national model for Medicaid service delivery by the federal government, including HRSA and HCFA. This protocol represents a component of that evaluation,from the patients' perspective.This study is being conducted in collaboration with the New York State Department of Health (NYSDOH) AIDS Institute. As a component of their Quality Management and Improvement Programs, Special Need Plans have agreed to assist with recruitment of participants to this evaluation. We will recruit 120 patients sampled from each of the six plans and follow these patients for initially a year with a possibility of continuing to interview them for up to two years. We will also recruit a sample of 360 current Medicaid fee for service patients to serve as comparison group. This sampling strategy will allow us to examine experiences in care and outcomes for different subgroups of patients within the plans, distinguish the affects of service differences among the plans and compare different plan enrollees to similar patients who remain in the Medicaid FFS program. Our longitudinal design will also permit us to examine prospective influences on comparison group patients' decisions to switch their coverage from Medicaid FFS to Special Needs Plans.

ELIGIBILITY:
Inclusion Criteria:

PWHA must meet the following criteria:

* Medicaid Special Needs Plans or Fee For Service as health insurance at the timeof enrollment;
* Age 18 years or older
* A current resident of New York State
* Able to respond to interview questions in English or Spanish.
* Express willingness and ability to complete a series of one-hour long interviews (interviews may be completed over two telephone sessions, if PWHAs prefer)
* Have cognitive and physical capacity to comprehend and complete the informed consent

Exclusion Criteria:

* Enrollment onto the study at an earlier site (we may encounter the same PWHA at more than one FFS recruitment site) • Staff members from Special Needs Plans or FFS Recruitment site determine that it is inadvisable to refer a PWHA to this study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The NYSDOH AIDS Institute will obtain Case Report Forms from Special Need Plans. and if they have agreed to receive mail and/or telephone calls regarding the plan they have signed up for. All patients will be informed at the time they join a Special Needs Plan that they may be contacted by evaluators working with the NYSDOH AIDS Institute who willwant to ask them about enrollment and care in the plan. Patients who have not agreed to receive mail will only be contacted by telephone.At this time, a call will be made to conduct screening using the Enrollment module and ask the selected Special Needs Plan patient about their willingness toparticipate in the study.
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2003-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
This study makes use of several new assessment approaches designed to provide a more in depth understanding of access to care, changes in care, and patient-reported outcomes. | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Rapkin, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Slaon-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer website — http://www.mskccc.org